CLINICAL TRIAL: NCT00771563
Title: Low Molecular Weight Heparin in Advanced Non Small Cell Lung Cancer (NSCLC): a Randomized Open Label Phase III Study Evaluating the Effect of Enoxaparin (Clexane) on Survival and Symptom Control in Patients With Stage IIIB and IV NSCLC Undergoing a Cisplatin Based First Line Chemotherapy: the SYRINGES Trial
Brief Title: Enoxaparin Low Molecular Weight Heparin (LMWH) in Advanced Non Small Cell Lung Cancer: Effect on Survival and Symptom Control in Patients Undergoing First Line Chemotherapy (SYRINGES)
Acronym: SYRINGES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Ethisch Comité UZ Antwerpen, Thoracale Oncologie Groep Antwerpen, University Hospital, Antwerp
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TOGA 0601; EudraCT 2007-007696-16
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; chemotherapy; Low Molecular Weight Heparin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Docetaxel; Enoxaparin; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Active Comparator): Chemotherapy without LMWH
  Interventions: Drug: cisplatin + docetaxel
- Arm B (Experimental): Chemotherapy with LMWH
  Interventions: Drug: cisplatin + docetaxel + enoxaparin

INTERVENTIONS:
Drug: cisplatin + docetaxel — docetaxel 75 mg/m2 d1 and cisplatin 75mg/m2 d1 (q 3wks for 4 cycles)
  Other Names: Platinol; Taxotere
  Arms: Arm A
Drug: cisplatin + docetaxel + enoxaparin — cisplatin 75 mg/m2 d1 and docetaxel 75 mg/m2 d1 (q 3 wks for 4 cycles) + daily enoxaparin 1mg/kg/d sc
  Other Names: Platinol; Taxotere; Clexane; LMWH
  Arms: Arm B

SUMMARY:
Rationale: a number of recent phase III randomized trials have shown a survival benefit of a treatment with subcutaneous low-molecular weight heparin in patients with advanced solid malignancies. The survival advantages observed in the studies persist for months after the active treatment with LMWHs. Therefore these survival advantages are thought to be due to effects of LMWHs on tumor cell biology.

First line treatment of advanced NSCLC patients with the Cisplatin + Docetaxel combination has been widely studied, and is amongst the most active treatments currently available. The occurrence of grade 3/4 thrombopenia in several phase III trials was in the 0-3% range, making it an ideal chemotherapy regimen to combine with LMWHs in the treatment of advanced NSCLC.

DETAILED DESCRIPTION:
Purpose: the aim of this study is to evaluate the potential beneficial antitumoral effect of LMWH enoxaparin in patients with locally advanced or metastatic NSCLC determined by the time to progression, the overall survival and the symptom control. LMWH will be added to a first line cisplatin-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic NSCLC (stage IIIB or IV)
* Patients who are not candidates for radical combined modality treatments or high-dose radiation therapy
* At least one measurable lesion according to RECIST criteria
* Good performance status
* Adequate haematological, renal and liver function
* Written informed consent

Exclusion Criteria:

* Previous chemotherapy for NSCLC
* Brain metastasis
* History of cerebral haemorrhage, neurosurgery within 3 previous months or surgery within the past 6 months
* Indication for anticoagulant therapy, thrombolytic therapy or antiplatelet therapy for cardiovascular disease
* Concomitant therapy with an anti-angiogenesis agent
* Contra-indication for LMWH
* Life expectancy of < 3 months
* Serious concomitant systemic disease, uncontrolled arterial hypertension, active peptic ulcer or other condition which does not permit study treatment or follow-up required to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2008-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | during chemotherapy and follow-up

SECONDARY OUTCOMES:
Symptom control evaluated with the Lung Cancer Symptoms Scale (LCSS) | during chemotherapy and follow-up
Overall Survival | during chemotherapy and follow-up
Best Overall Response | during chemotherapy and follow-up
Incidence of total documented thromboembolic and hemorrhagic events | during chemotherapy and follow-up
Overall safety and tolerability | during chemotherapy and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Paul R Germonpre, MD PhD, Principal Investigator — Universiteit Antwerpen
Locations (2):
- Belgium (2):
  - University Hospital Antwerp, Edegem, Antwerp
  - Centre Hospitalier Universitaire Sart Tilman, Liège, Liège

REFERENCES:
- [Derived] Rutjes AW, Porreca E, Candeloro M, Valeriani E, Di Nisio M. Primary prophylaxis for venous thromboembolism in ambulatory cancer patients receiving chemotherapy. Cochrane Database Syst Rev. 2020 Dec 18;12(12):CD008500. doi: 10.1002/14651858.CD008500.pub5. PMID 33337539